CLINICAL TRIAL: NCT07395258
Title: Phase I Open-label Dose Escalation Trial of BI 3923948 Monotherapy and in Combination With an Anti-PD-1 mAb in Patients With Advanced, Unresectable and/or Metastatic Solid Tumors
Brief Title: A Study to Test Different Doses of BI 3923948 Alone and in Combination With an Anti-PD-1 Antibody in People With Different Types of Advanced Cancer (Solid Tumors)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1538-0001; U1111-1319-8046 (Registry Identifier: WHO - International Clinical Trials Registry Platform (ICTRP)); 2025-521438-27-00 (EU CTIS Number)
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: BI 3923948 monotherapy (Experimental)
  Interventions: Drug: BI 3923948
- Arm B: BI 3923948 in combination with ezabenlimab (Experimental)
  Interventions: Drug: BI 3923948; Drug: Ezabenlimab

INTERVENTIONS:
Drug: BI 3923948 — BI 3923948
Drug: Ezabenlimab — Ezabenlimab
  Arms: Arm B: BI 3923948 in combination with ezabenlimab

SUMMARY:
This study is open to adults aged 18 and over or above legal age with different types of recurrent advanced cancer (solid tumors) that have spread to other parts of the body and that are accessible for injection and biopsy. This is a study for people for whom previous treatment was not successful or no treatment exists, with a life expectancy of at least 3 months after starting study treatment. The purpose of this study is to find the highest dose of a medicine called BI 3923948, that people with advanced cancer can tolerate, when taken alone and together with a type of antibody called a checkpoint inhibitor (anti-programmed cell death protein 1 antibody). Another purpose is to check whether the study treatment can fight cancer. In this study, BI 3923948 is given to people for the first time.

This study has 2 arms. In Arm A, participants get BI 3923948 alone for up to 3 months. In Arm B, participants get BI 3923948 in combination with a checkpoint inhibitor. Participants who take the combination treatment get BI 3923948 for up to 3 months and a checkpoint inhibitor for up to 1 year. BI 3923948 is given as injection(s) into the tumor, and the checkpoint inhibitor is given as an infusion into a vein. Participants get the medicines about every 3 weeks. This is called a treatment cycle. Only in treatment cycle 1 will participants get BI 3923948 twice in the first week.

Participants visit the site study site regularly. The number of study visits vary based on the study arm and treatment response. Some visits include an overnight stay. The doctors regularly check the participants' health and monitor the tumors. The doctors closely check the health of the participants and also take note of any health problems that could have been caused by the study treatment.

ELIGIBILITY:
Inclusion criteria:

1. Measurable disease as defined per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
2. Patient has 1 or more accessible lesions (2 or more preferred)
3. Eastern Cooperative Oncology Group (ECOG) score of 0 or 1
4. Life expectancy of at least ≥3 months after the start of the treatment according to the investigator's judgement Further inclusion criteria apply.

Exclusion criteria:

1. Patients with known primary brain tumors, leptomeningeal disease or untreated brain metastases. Subjects with previously treated brain metastases may participate provided the brain metastases are stable
2. Previous treatment with vesicular stomatitis virus (VSV)-based agents
3. Concomitant medication or condition considered a high risk for complications from injection
4. History of common terminology criteria for adverse events (CTCAE) v5 grade 3 or higher severe hypersensitivity reactions to previous anti-programmed cell death 1 (anti-PD-1)/anti-programmed cell death ligand 1 (PD-L1) monoclonal antibody (mAb) (Arm B only) Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03-10 (Estimated); Primary Completion 2028-02-20 (Estimated); Study Completion 2032-02-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Dose-limiting toxicities (DLTs) during the primary DLT evaluation period | up to 3 weeks

SECONDARY OUTCOMES:
Occurrence of DLTs during the on-treatment period | up to 12 months
Occurrence of Adverse Events (AEs) during the on-treatment period | up to 12 months

CONTACTS AND LOCATIONS:
Locations (10):
- United States (4):
  - Indiana University, Indianapolis, Indiana
  - University of Minnesota, Minneapolis, Minnesota
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- France (2):
  - CTR Leon Berard, Lyon
  - INS Gustave Roussy, Villejuif
- Universitätsklinikum Heidelberg, Heidelberg, Germany
- Spain (2):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Clinico De Valencia (INCLIVA), Valencia
- Karolinska Universitetssjukhuset Stockholm, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com